CLINICAL TRIAL: NCT05258604
Title: Endoscopic Band Ligation Versus Argon Plasma Coagulation in Management of Gastric Antral Vascular Ectasia; Randomized Clinical Trial
Brief Title: Endoscopic Band Ligation Vs APC in Management of GAVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Yousef Mohammed, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: endoscopic management of GAVE
Record Dates: First submitted 2022-01-21; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: GAVE - Gastric Antral Vascular Ectasia
MeSH Terms: conditions — Gastric Antral Vascular Ectasia | interventions — Argon Plasma Coagulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- argon plasma coagulation (APC). (Experimental): APC Standard APC equipment will be used, consisting of a high-frequency electrosurgical generator (ICC 350; ERBE, Tübingen, Germany), an argon source which is regulated automatically (APC 300) and APC probe.
  Interventions: Procedure: argon plasma coagulation
- endoscopic band ligation. (Experimental): endoscopic band ligation will be carried out using a Saeed Multi-Band Ligator (Cook Medical, WinstonSalem, NC), and ligation bands were placed on the GAVE.
  Interventions: Procedure: endoscopic band ligation

INTERVENTIONS:
Procedure: argon plasma coagulation — APC Standard APC equipment will be used, consisting of a high-frequency electrosurgical generator (ICC 350; ERBE, Tübingen, Germany), an argon source which is regulated automatically (APC 300) and APC probe.
  Arms: argon plasma coagulation (APC).
Procedure: endoscopic band ligation — endoscopic band ligation will be carried out using a Saeed Multi-Band Ligator (Cook Medical, WinstonSalem, NC), and ligation bands were placed on the GAVE.
  Arms: endoscopic band ligation.

SUMMARY:
* overall aim: To compare the efficacy and safety of endoscopic band ligation and endoscopic argon plasma coagulation for the management of gastric antral vascular ectasia.
* Secondary aims:

  1. Study risk factors of GAVE.
  2. Prevalence of GAVE among causes of non-variceal gastrointestinal bleeding.

DETAILED DESCRIPTION:
Gastric antral vascular ectasia (GAVE) is a capillary-type vascular malformation characterized endoscopically by red, angiomatous lesions originating in the antrum and organized either in stripes or in a diffuse pattern.

GAVE may cause chronic iron-deficiency anemia with or without the presence of overt gastrointestinal bleeding, manifested commonly by melena, may account for about 4% of the causes of non-variceal bleeding.

GAVE can be isolated or associated with systemic conditions, especially in patients with liver cirrhosis, scleroderma, chronic renal failure, and after bone marrow transplantation.

Multiple mechanisms have been proposed as the origin of its development. These have included gastric dysmotility leading to chronic mucosal trauma and subsequent fibromuscular hyperplasia and vascular ectasia or an autoimmune reaction to gastric blood vessels among the main contributing factors.

Management of GAVE-related gastrointestinal bleeding is a clinically challenging issue. In the last two decades, many therapeutic options and modalities have been applied for GAVE including medical, endoscopic, and surgical management.

Endoscopic management including different options such as cryotherapy, argon photo coagulation (APC), Neodymium-yttrium-aluminum garnet laser coagulation, radiofrequency ablation and endoscopic band ligation.

The first case using endoscopic band ligation as salvage treatment for GAVE was reported in 2006. After two sessions of EBL with a Multi-Band Ligature, hemoglobin became stable and serum ferritin normalized in 16 months of follow up.

Some studies show that management of GAVE with endoscopic band ligation superior to APC in bleeding cessation and fewer treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* • Both sexes will be included.

  * Age above 18 years old patients will be included.
  * With overt or occult bleeding from GAVE.
  * Characteristic endoscopic findings of GAVE: GAVE was limited to the antrum and its appearance either watermelon stomach or diffuse pattern.

Exclusion Criteria:

* • All causes of emergence upper GIT bleeding other than GAVE.

  * Patient with contraindication to general anesthesia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
prevalence of gastric antral vascular ectasia (GAVE) among other causes of gastrointestinal bleeding and study different endoscopic modalities in GAVE management according to its side effects and capacity in management of GAVE | two years
  prevalence OF GAVE will be assessed according to number of cases presented by gastrointestinal bleeding diagnosed as GAVE by upper endoscopy
  side effects of endoscopic modalities will be assessed according
  1. incidence of re-bleeding
  2. Need for blood transfusion according to numbers of packed red blood cells units.
  3. Hospital stay and total cost.
  4. post procedure gastric ulceration detected by upper endoscopy.

REFERENCES:
- [Background] Zepeda-Gomez S. Endoscopic Treatment for Gastric Antral Vascular Ectasia: Current Options. GE Port J Gastroenterol. 2017 Jul;24(4):176-182. doi: 10.1159/000453271. Epub 2016 Dec 21. PMID 29255747
- [Background] Fuccio L, Mussetto A, Laterza L, Eusebi LH, Bazzoli F. Diagnosis and management of gastric antral vascular ectasia. World J Gastrointest Endosc. 2013 Jan 16;5(1):6-13. doi: 10.4253/wjge.v5.i1.6. PMID 23330048
- [Background] Hung EW, Mayes MD, Sharif R, Assassi S, Machicao VI, Hosing C, St Clair EW, Furst DE, Khanna D, Forman S, Mineishi S, Phillips K, Seibold JR, Bredeson C, Csuka ME, Nash RA, Wener MH, Simms R, Ballen K, Leclercq S, Storek J, Goldmuntz E, Welch B, Keyes-Elstein L, Castina S, Crofford LJ, Mcsweeney P, Sullivan KM. Gastric antral vascular ectasia and its clinical correlates in patients with early diffuse systemic sclerosis in the SCOT trial. J Rheumatol. 2013 Apr;40(4):455-60. doi: 10.3899/jrheum.121087. Epub 2013 Feb 15. PMID 23418384
- [Background] Hsu WH, Wang YK, Hsieh MS, Kuo FC, Wu MC, Shih HY, Wu IC, Yu FJ, Hu HM, Su YC, Wu DC. Insights into the management of gastric antral vascular ectasia (watermelon stomach). Therap Adv Gastroenterol. 2018 Jan 14;11:1756283X17747471. doi: 10.1177/1756283X17747471. eCollection 2018. PMID 29399041
- [Background] Kantsevoy SV, Cruz-Correa MR, Vaughn CA, Jagannath SB, Pasricha PJ, Kalloo AN. Endoscopic cryotherapy for the treatment of bleeding mucosal vascular lesions of the GI tract: a pilot study. Gastrointest Endosc. 2003 Mar;57(3):403-6. doi: 10.1067/mge.2003.115. PMID 12612530
- [Background] American Society for Gastrointestinal Endoscopy Technology Committee. Mucosal ablation devices. Gastrointest Endosc. 2008 Dec;68(6):1031-42. doi: 10.1016/j.gie.2008.06.018. No abstract available. PMID 19028211
- [Background] Sinha SK, Udawat HP, Varma S, Lal A, Rana SS, Bhasin DK. Watermelon stomach treated with endoscopic band ligation. Gastrointest Endosc. 2006 Dec;64(6):1028-31. doi: 10.1016/j.gie.2006.05.006. Epub 2006 Aug 22. No abstract available. PMID 17140926
- [Background] Keohane J, Berro W, Harewood GC, Murray FE, Patchett SE. Band ligation of gastric antral vascular ectasia is a safe and effective endoscopic treatment. Dig Endosc. 2013 Jul;25(4):392-6. doi: 10.1111/j.1443-1661.2012.01410.x. Epub 2012 Dec 17. PMID 23808945
- [Background] Sato T, Yamazaki K, Akaike J. Endoscopic band ligation versus argon plasma coagulation for gastric antral vascular ectasia associated with liver diseases. Dig Endosc. 2012 Jul;24(4):237-42. doi: 10.1111/j.1443-1661.2011.01221.x. Epub 2011 Dec 29. PMID 22725108